CLINICAL TRIAL: NCT01355016
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of Inhaled MDT-637 in Healthy Volunteers
Brief Title: A Trial to Assess the Safety, Tolerability, and Pharmacokinetics of MDT-637 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MicroDose Therapeutx, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDT-637-CP-101
Record Dates: First submitted 2011-05-11; First posted 2011-05-17 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Drug Safety; Respiratory Syncytial Virus Infections
Keywords: RSV
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — VP-14637

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- MDT-637 (Experimental): Active formulation
  Interventions: Drug: MDT-637
- Placebo (Placebo Comparator): Matched Placebo Comparator
  Interventions: Drug: MDT-637

INTERVENTIONS:
Drug: MDT-637 — Inhaled doses of MDT-637 over a 24 hour period

SUMMARY:
The purpose of this study is to determine the range of single inhaled doses of a new dry powder product, MDT-637, that are safe and well-tolerated. This includes monitoring effects on pulmonary function and determination of blood levels of MDT-637 following inhalation.

ELIGIBILITY:
Inclusion Criteria:

* Males and/or surgically sterile or post-menopausal females (confirmed by FSH test); males must agree to practice barrier contraception until they are discharged from the study
* Willing to give written informed consent
* 18 to 50 years of age
* BMI of 19-30 Kg/m2
* Non-smoker (for at least 90 days prior to screening) and willing to abstain from smoking during the course of the study
* Good general health as determined by medical history, physical examination, ECG and clinical laboratory tests
* Willing to abstain from alcohol, caffeine, and xanthine-containing beverages for 24 hours prior to and 24 hours after dosing

Exclusion Criteria:

* Uncontrolled, clinically significant disease which in the opinion of the Principal Investigator and MDT would place the subject at risk through study participation or would confound the assessment of the safety of MDT-637
* Evidence of current or history of respiratory disease, including asthma, emphysema, chronic bronchitis, or cystic fibrosis
* History of significant nasal irritation from nasal inhalation of medication
* History of malignancy
* History of clinically significant alcohol or drug abuse
* Positive drug screen for drugs of abuse
* Positive test for HIV, Hepatitis B or Hepatitis C
* Allergy to lactose, or lactose intolerance
* Use of prescription medication within 14 days of Visit 2 or over-the-counter preparations, including dietary and herbal supplements, within 5 days of Visit 2
* Positive serum pregnancy test at Visit 1
* Inability to perform reproducible spirometry
* Abnormal FEV1, FVC, or FEV1/FVC (FEV1and FVC < 85% of predicted and variability of <5% or FEV1/FVC ratio < 0.7)
* Abnormal QTc interval at Visit 1(>450 msec in males or > 470 msec in females)
* Significant blood donation (or testing) in previous 8 weeks

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of 6 escalating doses of MDT-637 dry powder inhalation in healthy volunteers | Up to 22 days (including 14 day screening period)
  Safety measurements include Clinical Laboratory Evaluations, Pulmonary Function Tests (Spirometry), ECG, Vital Signs, Physical Examination and Assessment of Adverse Events.

SECONDARY OUTCOMES:
Plasma pharmacokinetics for MDT-637 dry powder inhalation | Multiple plasma samples collected up to 24 hours post first dose
  Plasma samples will be measured to determine MDT-637 pharmacokinetics as defined by Cmax
Trough MDT-637 Nasal Concentration | 24 hours
  Determination of MDT-637 concentration following nasal wash
Plasma pharmacokinetics for MDT-637 dry powder inhalation | 24 hours
  Plasma samples will be measured to determine MDT-637 pharmacokinetics as defined by Tmax
Plasma pharmacokinetics of MDT-637 dry powder inhalation | 24 hours
  Plasma samples will be measured to determine MDT-637 pharmacokinetics as defined by AUC

CONTACTS AND LOCATIONS:
Locations (1):
- West Coast Clinical Trials, Cypress, California, United States

REFERENCES:
- See also: Development Program Information — http://mdtx.com/pipeline/proprietary-products/mdt-637/